CLINICAL TRIAL: NCT03323580
Title: Effects of Intraoperative Goal-directed Fluid Therapy (GDFT) on the Postoperative Brain Edema in Neurosurgical Patients With Malignant Supratentorial Gliomas
Brief Title: Effects of Intraoperative GDFT on the Postoperative Brain Edema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Yuming Peng, Ph.D.,M.D., Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2017-10-24
Record Dates: First submitted 2017-10-24; First posted 2017-10-27 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Fluid Therapy; Brain Edema; Brain Tumor
MeSH Terms: conditions — Brain Edema; Brain Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GDFT group (Experimental): The patients will receive fluid therapy under goal directed.
  Interventions: Other: GDFT
- Routine group (Sham Comparator): The patients will receive routine fluid therapy.
  Interventions: Other: traditional fluid therapy

INTERVENTIONS:
Other: GDFT — Target parameter will be titrated with fluid bolus, and thus individual amount varied depending on the parameter value at that time. Maintenance of oxygenation, hemoglobin, blood glucose, core temperature and hemodynamics, such as mean arterial pressure and heart rate, will be applied according to the same standard for each patient.
  Arms: GDFT group
Other: traditional fluid therapy — Fluid therapy will be done without goal directed. Maintenance of oxygenation, hemoglobin, blood glucose, core temperature and hemodynamics, such as mean arterial pressure and heart rate, will be applied according to the same standard for each patient.
  Arms: Routine group

SUMMARY:
Whether a fluid protocol aiming for protecting vital organ perfusion or fluid restriction is favorable to post-craniotomy outcomes such as brain edema remains uncertain. To our knowledge, there has been no extensive and quantitative analysis of brain edema following SVV-based GDFT in neurosurgical patients with malignant supratentorial glioma. So the study aims to observe the effect of the stroke volume variation-based GDFT on the postoperative brain edema and decrease the incidence of postoperative complications in neurosurgical patients with malignant supratentorial gliomas.

ELIGIBILITY:
Inclusion Criteria:

1. Preoperative brain image indicating high-grade glioma (HGG), verified by postoperative histology of the World Health Organization (WHO) as grade III or IV tumors.
2. Age 18-65 years, and American Society of Anaesthesiologists (ASA) physical status I to III.
3. Signed informed consent.

Exclusion Criteria:

1. Renal insufficiency or the creatinine clearance is < 30 mL/kg.
2. Heart disease, New York Heart Association Functional Classification (NYHA) class II or higher heart failure, or if their cardiac ejection fraction is < 20%.
3. Chronic obstructive pulmonary disease.
4. Extensive peripheral arterial occlusive disease.
5. Coagulopathy.
6. Surgery in the prone position.
7. Recurrent carcinoma or tumor in the brain ventricular.
8. Body Mass Index <18.5 kg·m-2 or >30.0 kg·m-2.
9. Awake craniotomy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Actual)
Dates: Start 2018-11-26 (Actual); Primary Completion 2022-09-21 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Quantitative analysis of brain edema | Within 24 hours postoperatively
  Postoperative brain edema is defined as edema surrounding the surgical resection cavity, which will be evaluated through CT images.Image evaluators will manually delineate region of interest (ROI) and operative cavity on each slice. The area will be calculated automatically by PACS system. The total volume will be acquired by multiplying area and slice thickness. The volume of edema will be calculated by the totoal volume of edema plus cavity minus the volume of cavity.

SECONDARY OUTCOMES:
The incidence of delirium | During the first 3 postoperative days
  Delirium was assessed twice daily (between 8-10 am and between 6-8 pm) with the Confusion Assessment Method for Intensive Care Unit (CAM-ICU) for critical care patients, or the 3-minute Diagnostic interview for Confusion Assessment Method (3D-CAM) for ward assessments, combined with the Richmond Agitation Sedation Scale (RASS). Delirium assessments were only conducted in patients with RASS sedation score exceeding -4.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Liu X, Zhang X, Fan Y, Li S, Peng Y. Effect of intraoperative goal-directed fluid therapy on the postoperative brain edema in patients undergoing high-grade glioma resections: a study protocol of randomized control trial. Trials. 2022 Nov 19;23(1):950. doi: 10.1186/s13063-022-06859-9. PMID 36401274